CLINICAL TRIAL: NCT06765044
Title: Textbook Outcomes of Surgical Treatment of Acute Appendicitis
Brief Title: Textbook Outcomes in Urgent Appendectomy
Acronym: APPX_TEXTBOOK
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, Ana María González Castillo, Principal Investigator, Hospital del Mar
Other Study IDs: Appendicitis Textbook Outomes; CEIm number (Other: Hospital del Mar)
Record Dates: First submitted 2024-12-17; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Valid MeSH Conditions
Keywords: Textbook Outcomes; Laparoscopy; Acute Appendicitis; Open Surgery; Urgent Appendectomy
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A "textbook outcome" patient is defined as one whose surgical course is uneventful, with no complications, readmissions, or mortality. There is a lack of published research regarding textbook outcomes with an acute appendicitis that are treated with an appendectomy.

DETAILED DESCRIPTION:
The objective of this study is to analyze the attainment of textbook outcomes (TO) in patients undergoing urgent appendicectomy (UA) for acute appendicitis and to identify the factors associated with achieving TO.

ELIGIBILITY:
Inclusion Criteria:

* Acute Appendicits in older than 18 years old
* Acute Appendicitis that needs appendectomy

Exclusion Criteria:

* Age under 18 years old
* Other diagnostic than an Acute Appendicitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the admissions with diagnostic of Acute Appendicitis in an University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
Textbook Outcomes | 2022-2024
  Classical assessments, focused solely on mortality and morbidity, are increasingly considered insufficient. A more comprehensive approach, using composite measures, offers a more accurate evaluation, providing a multidimensional view and patient-centred healthcare appraisal. The textbook outcome (TO) is the most used objective composite measure to compare surgical quality across centres

SECONDARY OUTCOMES:
Appendectomy in less than 24h | 2022-2024
  From diagnostic of Acute Appendicitus to Surgical Treatment should be less than 24h
Hospital Stay less than 5 days | 2022-2024
  Optimal hospital stay should be less than 5 days
Intraoperative incidences | 2022-2024
  Intraoperative bleeding, perforation of the appendix, iatrogenic injury to other structures
Short antibiotics treatment | 2022-2024
  Less than 72h of antibiotic treatment
Patient comorbidities | 2022-2024
  Charlson Comorbidity Index
Surgical Risk | 2022-2024
  ASA Scoring System
Intraoperative appendicitis gradding | 2022-2024
  AAST classification AAST I: Acutely inflamed appendix, intact. AAST II:Gangrenous appendix, intact AAST III:Above, with evidence of local contamination AAST IV:Above, with abscess or phlegmon in region of appendix AAST V:Above, with addition of generalized purulent contamination away from appendix
  WSES Classification:
  Grade- 0 (normal looking) Grade-1 (inflamed) Grade- 2A and 2B (necrosis) Grade- 3A - 3B - 3C (perforated - inflammatory tumor) Grade- 4 (perforate - diffuse peritonitis)
Postperative complications | 2022-2024
  Clavien Dindo and CCI (https://www.cci-calculator.com/)
  Grade I: Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic, and radiological interventions.
  Grade II:Requiring pharmacological treatment with drugs other than such allowed for Grade I Grade III:Requiring surgical, endoscopic or radiological intervention. Grade IV:Life-threatening complication (including CNS complications)* requiring IC/ICU-management with single or multiorgan disfunction.
  Grade V: Death of a patient
Readmision index | 2022-2024
  Percentage of readmission

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 2025-2026